CLINICAL TRIAL: NCT04291729
Title: An Open Clinical Trial to Evaluate Ganovo（Danoprevir ） Combined With Ritonavir in the Treatment of SARS-CoV-2 Infection
Brief Title: Evaluation of Ganovo （Danoprevir ） Combined With Ritonavir in the Treatment of SARS-CoV-2 Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Ninth Hospital of Nanchang (Other)
Collaborators: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASC-CTP-NC-01
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ganovo+ritonavir with or without interferon nebulization (Experimental)
  Interventions: Drug: Ganovo+ritonavir+/-Interferon nebulization

INTERVENTIONS:
Drug: Ganovo+ritonavir+/-Interferon nebulization — Ganovo one tablet (100mg / tablet) at a time, twice a day, up to 14 days. Ritonavir one tablet(100mg / tablet) at a time, twice a day, up to 14 days.With or without spray inhalation of interferon, 50μg / time for adults, twice a day up to 14 days.

SUMMARY:
Evaluation of the efficacy and safety of Ganovo combined with ritonavir for patients infected with SARS-CoV-2.

DETAILED DESCRIPTION:
Given no specific antiviral therapies for new coronavirus pneumonia approved yet and Ganovo, an oral Hepatitis C virus protease inhibitor, approved in China in June 2018 , this open, controlled trial will evaluate the efficacy and safety of Ganovo in hospitalized patients infected with SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years old;
* Pneumonia patients with new coronavirus infection were confirmed to be positive by RT-PCR and clinical manifestations. The diagnosis standard refers to the diagnosis and treatment plan for pneumonia with new coronavirus infection (Current Trial Version);
* Patients with newly diagnosed respiratory system discomfort who have been hospitalized (the diagnosis time of respiratory system discomfort shall not exceed 7 days);
* Women and their partners who have no planned pregnancy for nearly half a year and are willing to take effective contraceptive measures within 30 days from the first administration of the study drug to the last administration;
* Agree not to participate in other clinical research within 30 days from the first administration of the study drug to the last administration;
* Patients who voluntarily sign informed consent.

Exclusion Criteria:

* The pneumonia patients with severe new coronavirus infection met one of the following conditions: respiratory distress, RR >= 30 times / min; or SaO2 / SpO2 <93% in resting state; or arterial partial pressure of oxygen (PaO2) / concentration of oxygen (FiO2) <300MMHG (1mmhg = 0.133kpa);
* Pneumonia patients with severe new coronavirus infection meet one of the following conditions: respiratory failure and need mechanical ventilation; or shock; or other organ failure combined with ICU monitoring treatment;
* Severe liver disease (such as child Pugh score >=C, AST > 5 times upper limit);
* Patients with contraindications specified in the instructions of ritonavir tablets;
* The pregnancy test of female subjects in the screening period was positive;
* The researchers judged that it was not suitable to participate in this clinical trial (for example, patients who may be transferred to another hospital during the study period; patients with multiple basic diseases, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Rate of composite adverse outcomes | 14 days
  Defined as SPO2≤ 93% without oxygen supplementation, PaO2/FiO2 ≤300mmHg or a respiratory rate ≥30 breaths per min without supplemental oxygen

SECONDARY OUTCOMES:
Time to recovery | 14 days
  Clinical recovery was defined as sustained (48 hours) alleviation of illness based on symptom scores (fever, cough, diarrhea, myalgia, dyspnea) all being absent and no evidence for progression (newly-presented dyspnea, SpO2 decline ≥3%, respiratory rate ≥ 24 breaths per min without supplemental oxygen).
Rate of no fever | 14 days
  Rate of no fever
Rate of no cough | 14 days
  Rate of no cough
Rate of no dyspnea | 14 days
  Rate of no dyspnea
Rate of no requiring supplemental oxygen | 14 days
  Rate of no requiring supplemental oxygen
Rate of undetectable New coronavirus pathogen nucleic acid | 14 days
  Rate of undetectable New coronavirus pathogen nucleic acid
Rate of mechanical ventilation | 14 days
  Rate of mechanical ventilation
Rate of ICU admission | 14 days
  Rate of ICU admission
Rate of serious adverse event | 14 days
  Rate of serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Yahong Chen, MD, Study Director — Ascletis Pharmaceuticals Co., Ltd.
Locations (1):
- The Ninth Hospital of Nanchang, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided